CLINICAL TRIAL: NCT03889392
Title: Evaluation of Nephrectomy Specimen to Verify a Mechanism of Intracranial Aneurysm Development in Autosomal Dominant Polycystic Kidney Disease Patients
Brief Title: Evaluation of Nephrectomy Specimen for Intracranial Aneurysm Development in ADPKD
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sung Shin, Associate Professor, Asan Medical Center
Other Study IDs: 2019-0310
Record Dates: First submitted 2019-03-18; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Kidney Transplant; Complications; Aneurysm, Brain; Polycystic Kidney Diseases
MeSH Terms: conditions — Intracranial Aneurysm; Polycystic Kidney Diseases | interventions — Kidney Transplantation; Nephrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — polycystic kidney specimen from nephrectomy operation during kidney transplantation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- polycystic kidney disease: Adult autosomal dominant polycystic kidney disease patients who received kidney transplantation at Asan Medical Center between 1994 and 2018
  Interventions: Procedure: Kidney transplantation and nephrectomy

INTERVENTIONS:
Procedure: Kidney transplantation and nephrectomy — Bilateral nephrectomy of polycystic kidneys are routinely performed during kidney transplantation in ADPKD patients

SUMMARY:
ADPKD is the most common form of hereditary kidney disease and is known to occur in 1 of 400 to 1000 population in the U.S. ADPKD consists of 2.8% of patients receiving kidney transplantation in the investigator's center. It is known that ADPKD is associated with vascular anomalies, including abdominal aneurysms, valvular anomalies and especially intracranial aneurysms. Intracranial aneurysms occur in 9~12% of the ADPKD population which is higher than 2~3% in the general population and is known to be associated with PKD1 or PKD2 heritage.

Until now, most of the studies regarding intracranial aneurysms in ADPKD are conducted in animal models, and there are only few cellular studies conducted from human samples. Total 154 patients received kidney transplantation for ADPKD from 1994 to December 2018 at Asan Medical Center, Seoul, Korea. While performing kidney transplantation to ESRD ADPKD patients, nephrectomy has been routinely performed for polycystic kidney and the nephrectomy specimens can be obtained. The objective of this study is to investigate the mechanism of intracranial aneurysm in ADPKD patients by analyzing gene characteristics from nephrectomy specimens.

DETAILED DESCRIPTION:
ADPKD is associated with PKD1 gene on chromosome 16 and PKD2 gene on chromosome 4 and these gene respectively code polycystin 1 and polycystin 2. Currently the hypotheses for increased intracranial aneurysm rate in ADPKD patients is that mutation of polycystin is not only confined to nephron tissues but also in endothelial cells and vascular smooth muscle cells and results in mutation of vascular phenotype. Also recent studies show polycystin complex causes cystic changes through mutation in primary cilia in renal epithelium. Wild type endothelial cells respond to fluid shear stress by regulating levels of intracellular calcium and nitric oxide, however, PKD1 or PKD2 mutation in fetal aortic endothelial cells revealed loss of these responses.

During kidney transplantation, bilateral nephrectomies are routinely performed to ADPKD patients. In this study, the investigators plan to perform PKD gene tests and gene sequencing from polycystic kidney nephrectomy specimens of154 ADPKD patients who received kidney transplantation at Asan Medical Center between 1994 and 2018. The aim of this study to analyze the gene mutation of ADPKD patients and investigate mechanisms associated with intracranial aneurysm occurence in ADPKD patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between age 18 and 80,
* Patients who received kidney transplantation for ADPKD at Asan Medical Center between 1994 and 2018,
* Patients who received nephrectomy for polycystic kidney

Exclusion Criteria:

* those who refuse or are unable to provide consent form,
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients between age 18 and 80, Patients who received kidney transplantation for ADPKD at Asan Medical Center between 1994 and 2018, Patients who received nephrectomy for polycystic kidney
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 1994-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Intracranial aneurysm | average of 5 years
  Occurrence of intracranial aneurysm

REFERENCES:
- [Background] Iglesias CG, Torres VE, Offord KP, Holley KE, Beard CM, Kurland LT. Epidemiology of adult polycystic kidney disease, Olmsted County, Minnesota: 1935-1980. Am J Kidney Dis. 1983 May;2(6):630-9. doi: 10.1016/s0272-6386(83)80044-4. PMID 6846334
- [Background] Collins AJ, Foley RN, Chavers B, Gilbertson D, Herzog C, Johansen K, Kasiske B, Kutner N, Liu J, St Peter W, Guo H, Gustafson S, Heubner B, Lamb K, Li S, Li S, Peng Y, Qiu Y, Roberts T, Skeans M, Snyder J, Solid C, Thompson B, Wang C, Weinhandl E, Zaun D, Arko C, Chen SC, Daniels F, Ebben J, Frazier E, Hanzlik C, Johnson R, Sheets D, Wang X, Forrest B, Constantini E, Everson S, Eggers P, Agodoa L. 'United States Renal Data System 2011 Annual Data Report: Atlas of chronic kidney disease & end-stage renal disease in the United States. Am J Kidney Dis. 2012 Jan;59(1 Suppl 1):A7, e1-420. doi: 10.1053/j.ajkd.2011.11.015. No abstract available. PMID 22177944
- [Background] Torres VE, Harris PC, Pirson Y. Autosomal dominant polycystic kidney disease. Lancet. 2007 Apr 14;369(9569):1287-1301. doi: 10.1016/S0140-6736(07)60601-1. PMID 17434405
- [Background] Ecder T, Schrier RW. Cardiovascular abnormalities in autosomal-dominant polycystic kidney disease. Nat Rev Nephrol. 2009 Apr;5(4):221-8. doi: 10.1038/nrneph.2009.13. PMID 19322187